CLINICAL TRIAL: NCT01199029
Title: An Open Label Study Evaluating The Effect Of Single Doses Of Pf-04308515 And Prednisone On Carbohydrate Metabolism Utilizing An Oral Glucose Tolerance Test In Healthy Adult Subjects
Brief Title: Single Dose Study Of PF-04308515 And Prednisone On Carbohydrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B0861004
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Healthy People; Glucocorticoids; Prednisone
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- (Part 1) 10 mg PF-04308515 (8hrs) (Experimental)
  Interventions: Drug: PF-04308515
- (Part 1) 10 mg PF-04308515 (12hrs) (Experimental)
  Interventions: Drug: PF-04308515
- (Part 1) 5 mg Prednisone (Active Comparator)
  Interventions: Drug: Prednisone
- (Part 2) X mg PF-04308515 (Experimental)
  Interventions: Drug: PF-04308515
- (Part 2) Y mg PF-04308515 (Experimental)
  Interventions: Drug: PF-04308515
- (Part 2) 5 mg Prednisone (Active Comparator)
  Interventions: Drug: Prednisone
- (Part 2) 20 mg Prednisone (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: PF-04308515 — 10 mg extemporaneous preparation of oral solution predosed 8 hours prior to Oral Glucose Tolerance Test(OGTT)
  Arms: (Part 1) 10 mg PF-04308515 (8hrs)
Drug: PF-04308515 — 10 mg extemporaneous preparation of oral solution predosed 12 hours prior to Oral Glucose Tolerance Test(OGTT)
  Arms: (Part 1) 10 mg PF-04308515 (12hrs)
Drug: Prednisone — 5 mg tablet predosed at 8 hours prior to Oral Glucose Tolerance Test (OGTT)
  Arms: (Part 1) 5 mg Prednisone
Drug: PF-04308515 — X mg of Pf-04308515 extemporaneous oral solution predosed at selected time from Part 1 prior to Oral Glucose Tolerance Test (OGTT)
  Arms: (Part 2) X mg PF-04308515
Drug: PF-04308515 — Y mg of Pf-04308515 extemporaneous oral solution predosed at selected time from Part 1 prior to Oral Glucose Tolerance Test (OGTT)
  Arms: (Part 2) Y mg PF-04308515
Drug: Prednisone — 5 mg tablet predosed at 8 hours prior to Oral Glucose Tolerance Test (OGTT)
  Arms: (Part 2) 5 mg Prednisone
Drug: Prednisone — 20 mg (5 mg tablets) predosed at 8 hours prior to Oral Glucose Tolerance Test (OGTT)
  Arms: (Part 2) 20 mg Prednisone

SUMMARY:
This study will investigate the effect of a single dose of PF-04308515 or prednisone on calculated measures of glucose tolerance and insulin resistance by using a modified oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* BMI 17.5 to 30.5 kg/m2 and total body weight >50 kg

Exclusion Criteria:

* Fasting glucose above the limits of the reference range for healthy individuals
* "No treatment" OGTT indicative of impaired fasting glucose or impaired glucose tolerance
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Fold change in AUC (0-4hr) relative to no treatment baseline for plasma glucose, plasma insulin and plasma C-peptide | 4 hours

SECONDARY OUTCOMES:
Pharmacodynamic effects on plasma glucose, plasma insulin, and plasma C-peptide | 3 days
Safety: adverse events, vital sign measurements, physical examination | 3 days
Pharmacokinetics: sparse PF-04308515 plasma samples will be collected | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kalamazoo, Michigan, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0861004&StudyName=Single%20Dose%20Study%20Of%20PF-04308515%20And%20Prednisone%20On%20Carbohydrate%20